CLINICAL TRIAL: NCT01019889
Title: Effect of Socheongryong-tang and Yeongyopaedok-san in Upper Respiratory Tract Infection
Acronym: ESYUI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Yang Chun Park, Professor, Korea Health Industry Development Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B070029
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Upper Respiratory Tract Infections
Keywords: upper respiratory tract infections; herbal medicine
MeSH Terms: conditions — Respiratory Tract Infections | interventions — sho-seiryu-to

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Experimental): Placebo (encapsulated starch + lactose)
  Interventions: Drug: Placebo
- SCRT(Socheongryong-tang ) (Experimental): encapsulated Socheongryong-tang extract
  Interventions: Drug: SCRT
- YPS (Yeongyopaedok-san) (Experimental): Encapsulated Yeongyopaedok-san extract
  Interventions: Drug: YPS

INTERVENTIONS:
Drug: SCRT — 4 capsules,three times daily, for 7days or within symptom disappearance
  Other Names: Xiao-qing-long-tang
  Arms: SCRT(Socheongryong-tang )
Drug: YPS — 4 capsules, three times daily, for 7days or within symptom disappearance
  Other Names: Lian-qiao-bai-du-san
  Arms: YPS (Yeongyopaedok-san)
Drug: Placebo — 4 capsules, three times daily, for 7days or within symptom disappearance
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Socheongryong-tang (SCRT) and Yeongyopaedok-san (YPS) are effective in the treatment of upper respiratory tract infection.

DETAILED DESCRIPTION:
Upper respiratory tract infections (URTIs) are the most prevalent disease of human beings, it incur a significant health burden on populations in terms of human suffering and economic losses. Usually, antibiotic therapy is not helpful since most infections are virally induced. Over 200 serologically different viral types are responsible for human URTIs, so that preventions of URTIs including vaccination are impassable. SCRT and YPS are widely used to treat the respiratory disease. The objective of this study is to determine the efficacy of SCRT and YPS in symptomatic relief of patients with URTIs.

ELIGIBILITY:
Inclusion Criteria:

* 18~60 years old
* Clinical diagnosis of common cold
* Occurring no longer than 48 hours before enrollment
* Presented with runny nose, sore throat, plugged nose, scratchy throat, cough, hoarseness, headache, muscle ache (runny nose, sore throat and at least 1 of others or 1 of runny nose, sore throat and at least 3 of others)

Exclusion Criteria:

* Allergic rhinitis, asthma, COPD, sinusitis (2 and more recurrence per year), septal deviation, anatomical otitis media, exudative pharyngitis
* Received antihistamines, NSAIDs, corticosteroids, antibiotics, decongestants
* Hepatic cancer, liver cirrhosis, renal failure, congestive heart failure
* Pregnant or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Changes of score daily measured by WURSS-K before, during and after treatment | daily (7 days)

SECONDARY OUTCOMES:
Time of symptom disappearance | daily
Changes of score daily measured by WURSS-K before, during and after treatment in pattern identification | daily (7days)

CONTACTS AND LOCATIONS:
Overall Officials: YangChun Park, Ph. D., Principal Investigator — Daejeon University